CLINICAL TRIAL: NCT06104878
Title: Effectiveness of A+AVD vs ABVD Regimens in Advanced Classical Hodgkin's Lymphoma Patients: A Retrospective, Multicentre, Medical Chart Review Study
Brief Title: A Study in Adults With Advanced Classical Hodgkin's Lymphoma (cHL) in Brazil Treated With Brentuximab Vedotin Together With Chemotherapy Compared to Chemotherapy Alone
Status: Withdrawn | Type: Observational
Why Stopped: Company decision after projects re-evaluation, taken before the study initiation
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brentuximab-5021
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABVD: Doxorubicin 25 mg/m^2 + Bleomycin 15 mg + Vinblastine 6 mg/m^2 + Dacarbazine 375 mg/m^2: Participants treated with doxorubicin 25 mg/m^2, bleomycin 15 mg, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 as first line therapy in each 28-day cycle for up to 6 cycles from July 1st, 2017, to December 31st, 2020, will be observed retrospectively.
  Interventions: Other: No Intervention
- A+AVD: Brentuximab Vedotin 1.2mg/kg+Doxorubicin 25mg/m^2 +Vinblastine 6mg/m^2 +Dacarbazine 375mg/m^2: Participants treated with brentuximab vedotin 1.2 mg/kg, doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 as first line therapy in each 28-day cycle for up to 6 cycles from July 1st, 2017, to December 31st, 2020, will be observed retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention will be administered in this study.

SUMMARY:
The main aim of this study conducted in Brazil is to understand if there is a difference in the length of time that Classical Hodgkin's Lymphoma (cHL) does not grow or spread further (also called progression free survival or PFS), and in the length of time that participants live with cHL if they are treated with Brentuximab Vedotin in combination with chemotherapy (A+AVD) or chemotherapy alone (ABVD).

A+AVD includes Brentuximab Vedotin + Doxorubicin + Vinblastine + Dacarbazine; ABVD includes Doxorubicin + Bleomycin + Vinblastine + Dacarbazine.

The study will be conducted by reviewing and collecting already existing medical records.

DETAILED DESCRIPTION:
This is an observational, multicenter and retrospective study to evaluate the effectiveness of A+AVD regimen compared to ABVD regimen as first-line therapy for the treatment of Brazilian participants with advanced cHL diagnosis.

The study will enroll approximately 200 participants who were treated with A+AVD or ABVD as first line therapy for at least one full cycle of 28 days, from July 1st, 2017, to December 31st, 2020. Participants will be identified from medical charts and will be assigned into following treatment groups:

* ABVD: Doxorubicin 25 milligrams per square meter (mg/m^2) + Bleomycin 15 milligram (mg) + Vinblastine 6 mg/m^2 + Dacarbazine 375 mg/m^2
* A+AVD: Brentuximab Vedotin 1.2 milligrams per kilogram (mg/kg) + Doxorubicin 25 mg/m^2 + Vinblastine 6 mg/m^2 + Dacarbazine 375 mg/m^2

This multi-center trial will be conducted in Brazil. The duration of the study will be 12 months. Participants will be followed up for at least 2 years after the last therapy cycle (treatment window considered for the study from July 1st, 2017, to December 31st, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced cHL (International Classification of Diseases and Related Health Problems 10th Revision [ICD-10] code C81.X). The diagnosis of cHL will be confirmed according to World Health Organization (WHO) classification. Advanced disease is defined as having the diagnosis at stage IIB, III or IV, based on Ann Arbor classification.
* Who received at least one full cycle of A+AVD or ABVD regimen as first-line treatment (first systemic therapy for cHL management; systemic therapy naïve participants) from July, 1st 2017 to December, 31st 2020; and who completed the 6-cycle treatment until the end of December 2020.
* At least 2 years of retrospective information from the index date (treatment window) and at least 2 years of follow-up (after the end of treatment).

Exclusion Criteria:

* With previous or concurrent malignancies, except participants with completely excised carcinoma in situ of any type and basal or squamous cell carcinoma of the skin.
* Who are simultaneously participating in another study.
* Who participated in the ECHELON-1 Clinical Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed of advanced cHL treated with A+AVD or ABVD as first-line systemic therapy in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From the index date (treatment start date) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first (up to 5.5 years)
  The PFS will be calculated as the time (months) from the index date to the first documentation of objective tumor progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From index date (treatment start date) to death by any cause during the study follow-up period (up to 5.5 years)
  The OS is defined as time from index date (treatment start date) to death by any cause during the study follow-up period.
Number of Participants Stratified by Vital Status on Last Follow up Visit | Up to approximately 5 years (Follow-up Period)
  Latest information about participants vital status (alive, death, lost of follow-up) will be reported.
Number of Deaths and Cause of Deaths | Up to approximately 5.5 years
  Number of deaths and different cause of deaths will be reported.
Time to Next Treatment (TTNT) | From the date of initiation of a treatment to the date of commencement of the next line of therapy (up to 5.5 years)
  The TTNT is defined as interval from the date of initiation of a treatment to the date of commencement of the next line of therapy.
Treatment-Free-Interval (TFI) | Up to approximately 5.5 years
  The TFI is defined as interval between the end of one regimen and the start of the next regimen (death or the end of follow-up are censoring events).
Number of Participants With Serious Adverse Events (SAEs) During Follow-up Period | Up to approximately 5 years (Follow-up Period)
  A SAE is defined as signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.
Number of Participants With Adverse Events (AEs) During follow-up Period | Up to approximately 5 years (Follow-up Period)
  An adverse event (AE) is any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product (including peripheral neuropathy and neutropenia).
Number of Participants With AEs Leading to Drug Discontinuation or Dose Reduction During Follow-up Period | Up to approximately 5 years (Follow-up Period)
  An AE is any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
Number of Participants With Most Common SAEs and Total AEs During Follow-up Period | Up to approximately 5 years (Follow-up Period)
  A SAE is defined as signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event. Most common SAEs are defined as most frequent SAEs occurred during the study. An AE is any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
Number of Treatment Cycles Participants Received | Up to approximately 6 months
  Number of treatment cycles received by participants will be reported. The length of each treatment cycle will be 28 days.
Percentage of Participants With Completed Treatment Cycles | Up to approximately 6 months
  Participant who completed 6 cycles of treatment during the treatment window (July 1, 2017, to December 31, 2020) will be considered completed. The length of each treatment cycle will be 28 days.
Number of Participants With Treatment Interruption and Main Reasons | Up to approximately 6 months
  Number of participant's that interrupted their treatment and the main reason will be reported. Reasons includes economical (example, healthcare insurance issues, cost-related, access barriers, etc.), participant's decision, adverse event (including toxicity), diseases progression, medical decision, death, other.
Number of Participants With Comorbidities and Comorbidities per Type | Up to approximately 5.5 years
  Comorbidities may include diabetes, obesity, autoimmune disease (example, arthritis, lupus and others), infectious disease (example, human immunodeficiency virus, Epstein Barr virus), cardiovascular disease (example, congestive heart failure, rhythm abnormalities, hypertension), dyslipidemia, cerebrovascular disease, gastrointestinal disease (example, gastritis, ulcer), pulmonary disease (example, chronic pulmonary disease, chronic obstructive disease), liver disease, renal disease, thyroid disease, depression, neurologic (example neuropathies), other cancers, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Brazil (6):
  - Hospital São Rafael - Instituto D'Or de Pesquisa e Ensino, Salvador, Estado de Bahia
  - Instituto D'Or de Pesquisa e Ensino, Brasília, Federal District
  - Oncoclinicas Rio de Janeiro S.A, Rio de Janeiro
  - Beneficência Portuguesa de São Paulo - Real Benemerita Associação Portuguesa de Beneficência, São Paulo
  - Hospital Alemão Oswaldo Cruz - HAOC, São Paulo
  - AC Camargo Cancer Center / Fundação Antonio Prudente Liberdade, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/875c87babb67426e?idFilter=%5B%22Brentuximab-5021%22%5D